CLINICAL TRIAL: NCT06449924
Title: An Endotracheal Tube Inserted to the Level of the Hypopharynx is an Easy, Safe, and Effective Technique for Ventilation of Pediatric Patients: A Prospective Observational Study
Brief Title: An Endotracheal Tube Inserted to the Level of the Hypopharynx
Status: Completed | Type: Observational
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Roland Kaddoum, Principal Investigator, American University of Beirut Medical Center
Other Study IDs: BIO-2024-0114
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Intubation; Difficult or Failed; Pediatric ALL; Ventilator Lung
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Endotracheal tube — Endotracheal Tube Inserted to the Level of the Hypopharynx

SUMMARY:
The goal of this observational study is to assess the incidence of successful ventilation using an ETT inserted orally above the vocal cords in pediatric patients undergoing surgeries. The main question it aims to answer are:

Is the use of an endotracheal tube (ETT), positioned in the hypopharynx with its tip placed just above the vocal cords an easy, safe and effective way for the ventilation of pediatric patients who are undergoing surgery under general anesthesia via orotracheal intubation?

The procedures to be performed in this study are standard of care. They are also used by pediatric anesthesiologists in the oral intubation of pediatric patients suffering from tumor or abscess.

DETAILED DESCRIPTION:
Background: Tracheal intubation can be challenging in the pediatric age group. The difficult airway algorithm is followed starting with ventilation via a facemask. In cases of difficulties in intubation and ventilation, and especially in neonates and small infants, oxygen desaturation can happen very quickly and can be life threatening. The endotracheal tube (ETT), which is readily available and bypasses the tongue of the patient, can provide a safe and efficient ventilation.

Specific Aim (s): In our study, we aim at assessing the incidence of successful ventilation using an ETT inserted orally above the vocal cords in pediatric patients undergoing surgeries. Secondary objectives include comparing the rate of successful ventilation between attending anesthesiologist and residents, assessing the incidence of success at first attempt, incidence of severe hypoxemia (SPO2 less than 85%), and incidence of adverse events such as bradycardia, stomach insufflation, laryngospasm, and desaturation.

Methods: This prospective observational study will include infants and children under 6 years of age who undergo surgeries at the American University of Beirut Medical Center (AUBMC). The tube will be inserted orally above the vocal cords following which ventilation will be attempted. The exclusion criteria include pediatric patients with an existing endotracheal tube, a BMI > 30 kg/m2, a risk of aspiration or a history of gastroesophageal reflux disease (GERD), and those undergoing emergency surgeries or whose legal guardian/representative is unwilling/unable to provide an written consent. The primary outcome is to assess successful ventilation (chest rise, end tidal CO2 wave and SpO2 levels).

Significance: This ETT technique is simple to implement and use, requiring no special training or equipment. This technique can save time by ensuring patients' oxygenation and ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children under 6 years of age undergoing surgery
* Legal guardian/representative willing to sign consent

Exclusion Criteria:

* Existing endotracheal tube
* BMI > 30 kg/m2
* Patient with a risk of aspiration of history of GERD
* Inability or unwillingness of research participant's legal guardian/ representative to give consent
* Need for emergency surgery
* ASA Ⅲ-Ⅳ
* Neonates below 28 days of age

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants and children under 6 years of age who undergo surgeries at the American University of Beirut Medical Center (AUBMC).
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Successful ventilation | During intubation
  Successful ventilation which is evaluated according to the following criteria:
  Delivery of tidal volume that makes the chest rise visibly, oxygen saturation by pulse oximeter not less than the value recorded after pre oxygenation and four end tidal CO2 waveforms.

SECONDARY OUTCOMES:
Rate of successful ventilation for attendings compared to that for residents | During intubation
  Rate of successful ventilation for attendings compared to that for residents
Incidence of success at first attempt | During intubation
  Incidence of success at first attempt
Incidence of severe hypoxemia | During intubation
  Incidence of severe hypoxemia (SPO2 less than 85%)
Incidence of adverse events | During intubation
  Incidence of adverse events such as bradycardia, stomach insufflation, laryngospasm, and desaturation

CONTACTS AND LOCATIONS:
Overall Officials: Roland Kaddoum, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No